CLINICAL TRIAL: NCT06858007
Title: Open, Non-comparative Study to Evaluate the Effectiveness and Safety of the Medical Device KOS® M in Lip Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Beauty Kozmetik (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGMQUA/0224/MD
Record Dates: First submitted 2025-02-04; First posted 2025-03-05 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lip Augmentation
Keywords: Lip augmentation improvement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOS® M (Other): An open, non-comparative, interventional single-armed clinical trial.
  Interventions: Device: KOS® M

INTERVENTIONS:
Device: KOS® M — Delivery of medical device as injection

SUMMARY:
The utilization of minimally invasive techniques has brought about a transformative shift in the approach to face rejuvenation, potentially representing one of the most notable advancements in facial plastic surgery in recent times. Originally employed to address the presence of fine lines and wrinkles, the application of fillers has now evolved to encompass the remediation of volume depletion and the enhancement of the aging visage.

Over a period of time, the convex shape of the midface region has the potential to undergo a flattening or concave transformation.

KOS® M in the dermis regulates water balance, osmotic pressure and ion flow and functions as a sieve, excluding certain molecules, enhancing the extracellular domain of cell surfaces and stabilizes skin structures by electrostatic interactions.

The Research Question of the present study is the following: to collect sufficient clinical data to demonstrate compliance with the General Safety and Performance Requirements of KOS® M when used as intended.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the subject
* Females and males ≥ 22 years of age
* Scoring 0 (minimal), 1 (mild) and 2 (moderate) on the 5-point Allergan LFS
* Have established a realistic treatment goal that the physician agrees is achievable, i.e., have realistic expectations of aesthetic results
* Ability to follow study instructions and likely to complete all required visits
* Reliable methods of contraception which result in a low failure rate (i.e. less than 1 % per year) for women of childbearing potential, e.g. implants, injectables, combined oral contraceptives, some intrauterine-devices, sexual abstinence or vasectomized partner) for the entire study duration.

Exclusion Criteria:

1. Has Inflamed or infected skin in or near the studied zones
2. History of or active autoimmune disease/immune deficiency
3. History of any disease resulting in changes of facial contour or edema of the face during the study period
4. Significant abnormalities of the lips
5. Has lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
6. Has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator
7. Has undergone oral surgery (e.g., tooth extraction, orthodontia, or implantation) within 6 weeks before enrollment or is planning to undergo any of these procedures during the study
8. Has ever undergone facial plastic surgery or received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
9. Has undergone semipermanent dermal filler treatment (e.g., calcium hydroxylapatite, poly-L- lactic acid) in the lower face (below the orbital rim) within 24 months before enrollment or is planning to undergo such treatment during the study
10. Has undergone temporary dermal filler treatment (e.g., hyaluronic acid or collagen) in the lower face (below the orbital rim) within 12 months before enrollment or is planning to undergo such treatment during the study
11. Taking medications and/or substances known to increase coagulation time (e.g., aspirin, ibuprofen, or herbal supplements) 10 days prior to treatment
12. Has undergone mesotherapy or cosmetic resurfacing (laser, photo-modulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) anywhere in the face or neck, or Botulinum toxin injections in the lower face (below the orbital rim) within 6 months before enrollment or is planning to undergo any of these procedures during the study
13. Prone to hypertrophic scars
14. History of allergy to hyaluronic acid or any of the product's components
15. History of allergy to lidocaine or local anaesthesia of amide compounds
16. Known case of porphyria
17. Pregnancy or lactation
18. Have a condition or be in a situation that, in the physician's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
19. Untreated epilepsy
20. Hypersensitivity to gram positive bacterial proteins as hyaluronic acid is produced by Streptococcus type bacteria.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of KOS® M in lip augmentation | 3 months
  The primary objective of the study is to evaluate the effectiveness of KOS® M in lip augmentation by assessing changes in the Allergan Lip Fullness Scale (ALFS). Response is defined as a ≥1 point improvement in ALFS at 3 months after last treatment.
  Allergan Lip Fullness Scale - from Minimal (Flat or nearly flat contour; minimal red lip shows) to Very Marked (Very significant red lip shows, lower lip pout, and lip pout)

SECONDARY OUTCOMES:
Effectiveness on KOS® M in lip augmentation | 3 months
  Effectiveness on KOS® M in lip augmentation through the assessment of the change in ALFS Allergan Lip Fullness Scale - from Minimal (Flat or nearly flat contour; minimal red lip shows) to Very Marked (Very significant red lip shows, lower lip pout, and lip pout)
Effectiveness on KOS® M in lip augmentation | 3 months
  Effectiveness on KOS® M in lip augmentation through the assessment of the change in FACE-Q Satisfaction with lips FACE-Q Satisfaction with lips - from 1 (Very Dissatisfied) to 4 (Very satisfied)
Effectiveness on KOS® M in lip augmentation | 3 months
  Effectiveness on KOS® M in lip augmentation through the assessment of the change in GAIS GAIS-The global aesthetic improvement scale - from 1 (very much improved) to 5 (worse)
Change in the ALFS (Allergan Lip Fullness Scale) Grade from baseline | 1, 3, 6 and 12 months
  Change in the ALFS (Allergan Lip Fullness Scale) Grade from baseline at 1, 3, 6 and 12 months after the last treatment.
  Allergan Lip Fullness Scale - grade from Minimal (Flat or nearly flat contour; minimal red lip shows) to Very Marked (Very significant red lip shows, lower lip pout, and lip pout)
Proportion of participants with at least 1-point improvement from baseline on the ALFS | 1,6 and 12 months
  Proportion of participants with at least 1-point improvement from baseline on the ALFS at 1,6 and 12 months after the last treatment (response rates) Allergan Lip Fullness Scale - grade from Minimal (Flat or nearly flat contour; minimal red lip shows) to Very Marked (Very significant red lip shows, lower lip pout, and lip pout)
Change from baseline in FACE-Q Satisfaction with Lips scores | 1, 3, 6 and 12 months
  Change from baseline in FACE-Q Satisfaction with Lips scores at 1, 3, 6 and 12 months after the last treatment.
  FACE-Q Satisfaction with Lips scores - from 1 (Very Dissatisfied) to 4 (Very satisfied)
Proportion of participants having a positive aesthetic evolution on the 5-point Global Aesthetic Improvement Scale (GAIS) | 1, 3, 6 and 12 months
  Proportion of participants having a positive aesthetic evolution on the 5-point Global Aesthetic Improvement Scale (GAIS) evaluated by the physician and subject on the lips at 1, 3, 6 and 12 months after the last treatment GAIS (The Global Aesthetic Improvement Scale) - from 1 (Very much improved) to 5 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Behnam D Bayatani, Study Chair
Locations (1):
- Clinica Beyond Dental, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attenello NH, Maas CS. Injectable fillers: review of material and properties. Facial Plast Surg. 2015 Feb;31(1):29-34. doi: 10.1055/s-0035-1544924. Epub 2015 Mar 12. PMID 25763894
- [Background] Werschler WP, Fagien S, Thomas J, Paradkar-Mitragotri D, Rotunda A, Beddingfield FC 3rd. Development and validation of a photographic scale for assessment of lip fullness. Aesthet Surg J. 2015 Mar;35(3):294-307. doi: 10.1093/asj/sju025. PMID 25805282
- [Background] Dayan S, Bruce S, Kilmer S, Dover JS, Downie JB, Taylor SC, Skorupa A, Murphy DK. Safety and Effectiveness of the Hyaluronic Acid Filler, HYC-24L, for Lip and Perioral Augmentation. Dermatol Surg. 2015 Dec;41 Suppl 1:S293-301. doi: 10.1097/DSS.0000000000000540. PMID 26618456